CLINICAL TRIAL: NCT06637345
Title: Identification of Prognostic and Predictive Biomarkers of Toxicity in Patients With Malignant Pleural Mesothelioma and Treated With High Doses of Radiotherapy (MESORTIBO)
Acronym: MESORTIBO
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-63
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Pleural Mesothelioma Malignant
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients treated with RT with radical intent from 01 January 2014 to the date of study approval
- Prospective cohort: Patients eligible for radical intent radiotherapy treatment radical, from the date of study approval

SUMMARY:
Malignant pleural mesothelioma (MPM) is a tumour that originates from the pleural layers (visceral and parietal) that envelop the lungs and the inner wall of the thoracic cage.

In other tumour contexts, numerous studies have demonstrated a synergistic effect between RT and Immune Checkpoint Inhibitors (ICIs), mainly due to immunogenic effects attributed to high doses of RT and ICIs-mediated activation of anti-tumour T lymphocytes.

Both treatments, RT and immunotherapy, have demonstrated a survival advantage in MPM, but are associated with non-negligible pulmonary toxicity. Therefore, the combination of these 2 therapeutic approaches requires a careful assessment of risk factors for the occurrence of toxicity. The identification of circulating biomarkers capable of predicting the onset of severe toxicity induced by radical radiation treatment is an important clinical need in MPM.

This study aims to monitor circulating biomarkers, such as molecules involved in inflammation and oxidative stress and cellular effectors modulated by radiation treatment and potentially associated with the development of toxicity and/or markers of an immunogenic effect of radiotherapy in the peripheral blood of subjects with malignant pleural mesothelioma for treatment with radical hemithoracic radiotherapy.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a tumour that originates from the pleural layers (visceral and parietal) that envelop the lungs and the inner wall of the thoracic cage.

In other tumour contexts, numerous studies have demonstrated a synergistic effect between RT and Immune Checkpoint Inhibitors (ICIs), mainly due to immunogenic effects attributed to high doses of RT and ICIs-mediated activation of anti-tumour T lymphocytes.

Both treatments, RT and immunotherapy, have demonstrated a survival advantage in MPM, but are associated with non-negligible pulmonary toxicity. Therefore, the combination of these 2 therapeutic approaches requires a careful assessment of risk factors for the occurrence of toxicity. The identification of circulating biomarkers capable of predicting the onset of severe toxicity induced by radical radiation treatment is an important clinical need in MPM.

This study aims to monitor circulating biomarkers, such as molecules involved in inflammation and oxidative stress and cellular effectors modulated by radiation treatment and potentially associated with the development of toxicity and/or markers of an immunogenic effect of radiotherapy in the peripheral blood of subjects with malignant pleural mesothelioma for treatment with radical hemithoracic radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age;
* Ability to understand, accept and sign consent informed;
* Histological diagnosis of malignant pleural mesothelioma;
* Previous administration of chemotherapy;
* Previous non-radical surgical approach (diagnostic thoracoscopy or R1-R2 surgery);
* Subject eligible for or already treated with RT on hemithorax for radical purposes (50 Gy in fractions on hemithorax + possible boost 60 Gy on residual PET+)

Exclusion Criteria:

* Disease not histologically established
* Progression pattern not amenable to radiation treatment (ipsilateral or metastatic intrathoracic extensive disease);
* Metastatic patient at diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-metastatic MPM previously treated with chemotherapy, undergoing a non-radical long-sparing surgical approach and treated with RT with radical intent (retrospective cohort) or eligible for RT with radical intent (prospective cohort)
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Association between biomarker levels measured at the end of radiation treatment and pulmonary toxicity of grade ≥2 associated with RT developed as an acute (within 6 months) or late (after 6 months) event | up to 36 months
  Differences in fold change of selected biomarkers, between subjects experiencing or not experiencing acute or late toxicity

SECONDARY OUTCOMES:
Relation between the severity of radio-induced toxicity and trend of biomarkers associated with it | up to 36 months
  Evaluation of linear trend of biomarkers fold change in relation with toxicity severity
Identifying biomarkers associated with lung toxicity potentially predictive of pulmonary fibrosis | up to 36 months
  Difference in frequencies of selected biomarkers between subgroups of patients with or without pulmonary fibrosis
Identifying signs of radio-induced immunomodulation among significant changes induced by hemithoracic radical radiotherapy in analysed biomarkers | up to 36 months
  difference in median values of selected biomarkers before and after treatment
Association between the levels of biomarkers measured at the end of treatment radiation and overall survival (OS) at 24 months | 24 moths after end of treatment
  Relation between overall survival and levels of biomarkers fold change using Cox regression. OS will be defined as time from beginning of the therapy until death from any cause or end of follow-up, whichever comes first.
To assess the prognostic potential of basal levels of analysed biomarkers | up to 36 months
  Relation between OS and pretreatment levels of selected biomarkers. Levels of biomarkers will be dichotomized based on pretreatment median value. Kaplan-Meier method and log rank test will be used. OS will be defined as time from beginning of the therapy until death from any cause or end of follow-up, whichever comes first.
Association between the levels of biomarkers variation (between baseline and treatment end) and Progression Free Survival (PFS) at 12 months | 12 months after end of treatment
  Relation between PFS and levels of biomarkers fold change compared to pre-treatment value. PFS will be defined as time from beginning of the therapy until objective PD, death or end of follow-up, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Revelant, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy